CLINICAL TRIAL: NCT00506272
Title: Inpatient Self Monitoring and Administration Study (ISMAS)
Acronym: ISMAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Atlanta VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Peter Thule, Chief, Section Endocrinology, Atlanta VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Emory IRB: 805-2006
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Diabetes Mellitus; Hyperglycemia; Hypoglycemia
Keywords: diabetes mellitus; hyperglycemia; hypoglycemia; self care
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia; Hypoglycemia | interventions — Blood Glucose Self-Monitoring; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard care (Experimental): Patients admitted for elective surgery will receive standard diabetes care, including but not limited to finger stick blood glucose determinations, and insulin injections delivered by the nursing staff.
  Interventions: Procedure: Standard care
- Patient administered care (Experimental): Patients will self-monitor and record finger-stick blood glucose measurements, and self administer insulin at doses agreed upon with the consulting endocrinology in-patient service.
  Interventions: Procedure: Self blood glucose monitoring and insulin administration

INTERVENTIONS:
Procedure: Self blood glucose monitoring and insulin administration — Patients will monitor blood glucose using a hand-held blood glucose monitor, and self-administer insulin
  Arms: Patient administered care
Procedure: Standard care — finger-stick blood glucose values to be obtained and all insulin administration to be delivered by nursing staff
  Arms: Standard care

SUMMARY:
ISMAS is designed to test the hypothesis that self management of insulin dependent diabetes mellitus by selected patients admitted for elective surgery is more efficacious than standard care with respect to overall glycemic control, attaining finger-stick blood sugars, and administering insulin.

ELIGIBILITY:
Inclusion criteria:

1. Male or female, age < 80
2. Most recent hemoglobin A1C within the past 6 months < 12%
3. Recent history of regular self-administered peripheral blood glucose checks as an outpatient
4. Recent history of insulin self-administration at least twice a day as an outpatient
5. Admitted for a hospitalization anticipated to last at least 3 days
6. Mini Mental Status Examination (MMSE) ≥ 25 at admission and the same or better post-operatively
7. All patients will be actively followed by the Endocrinology inpatient consultation team during the hospitalization.

Exclusion criteria:

1. Currently receiving peritoneal or hemodialysis
2. Patients with unstable angina
3. History of myocardial infarction within 3 weeks prior to enrollment
4. Current admission due to or associated with altered mental status or encephalopathy
5. History of an episode of altered mental status or encephalopathy within the 4 weeks prior to enrollment
6. A confirmed diagnosis of dementia
7. Inability to self-adjust insulin
8. No recent history of ability to perform regular peripheral blood glucose checks
9. Frequency of hypoglycemia (< 60 mg/dL) > twice/week by history
10. Inability to eat without assistance
11. Study objectives will not be pursued in patients during stays in any intensive care unit.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-12; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
number of blood glucose measurements obtained/number of blood glucose measurements ordered | patients will be followed for the duration of hospital stay, an expected average of 5 days
number of insulin doses administered/number of insulin doses prescribed | patients will be followed for the duration of hospital stay, an expected average of 5 days
average blood glucose | patients will be followed for the duration of hospital stay, an expected average of 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Thule, MD, Principal Investigator — Atlanta VA Medical Center
Locations (1):
- Atlanta VA Medical Center, Decatur, Georgia, United States